CLINICAL TRIAL: NCT04992975
Title: Brain Iron Toxicity and Neurodegeneration - An Ultrahigh Field (7T) MRI Study
Brief Title: Brain Iron Toxicity and Neurodegeneration - A 7T MRI Study
Acronym: BITaN
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19NS038
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-02

CONDITIONS: Prodromal Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Ultrahigh Field MRI; 7T MRI; QSM
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples will be stored and APOe status will be checked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alzheimer's disease: Patients with Early Onset Alzheimer's disease (with known cerebrospinal fluid Amyloid/tau status) during prodromal or mild phase will have MRI of the brain at 7T, neurocognitive assessments, and blood test to check APOe status.
  Repeat neuroimaging and neurocognitive tests after one year.
  Interventions: Other: MRI at 7T
- Control group: Age and gender matched individuals with normal cognition will have MRI of the brain at 7T, neurocognitive assessments and blood test to check APOe status.
  Repeat neuroimaging, neurocognitive tests after one year.
  Interventions: Other: MRI at 7T

INTERVENTIONS:
Other: MRI at 7T — MRI at 7T

SUMMARY:
A longitudinal observational neuroimaging study of individuals with Early Onset Alzheimer's disease during the prodromal phase, and matched control group - Ultrahigh Field MRI study at 7T

DETAILED DESCRIPTION:
This study aims to determine whether high resolution MRI at 7T and Quantitative Susceptibility Mapping (QSM) can demonstrate a specific pattern of iron overload in strategically important areas of brain as a sensitive marker of pathological Alzheimer's disease i.e. patients with subjective or mild cognitive impairment associated with Amyloid or tau pathological state in the cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Patients with pathological diagnosis of Alzheimer's disease according to the National Institute on Aging and Alzheimer's Association, NIA-AA, criteria (Alzheimer's group) or cognitively normal individuals within 1.5 standard deviation of normal in all tests (control group)

Exclusion Criteria:

* Lack of mental capacity to consent to study involvement
* Not speaking English before age 5 years
* Learning disability
* Schizophrenia
* Substance misuse
* Implanted devices not certified as compatible with ultra-high field MRI (e.g. cardiac pacemaker)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Alzheimer's Group: Preclinical or Prodromal Alzheimer's disease classified as either A+T-N- or A+T+N- Control Group: individual within 1.5 standard deviation of normal cognition in all tests
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Quantitative Susceptibility Mapping, QSM (from 7T MRI data) to hippocampal subfield volume loss at 1 year | one year
  Relationship between QSM at recruitment and to hippocampal subfield volume (QSM and hippocampal subfield volume are obtained from 7T MRI Susceptibility Weighted and T1 Weighted images)

SECONDARY OUTCOMES:
cross-sectional and longitudinal changes in QSM in the hippocampal subfields | one year
  cross-sectional and longitudinal changes in QSM in the local hippocampal subfield QSM and volume loss after 1 year. QSM and hippocampal subfields volume will be obtained from 7T MRI data
neuropsychological measures in relation to QSM and volume loss in hippocampal subfields | one year
  neuropsychological measures at 0 and 12 months in relation to QSM and volume loss in hippocampal subfields (adjusted for APOe). QSM and hippocampal subfield volume loss are obtained from 7T MRI Susceptibility Weighted and T1 Weighted images.

CONTACTS AND LOCATIONS:
Overall Officials: Akram Hosseini, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, East Midland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hari I, Adeyemi OF, Gowland P, Bowtell R, Mougin O, Vesey P, Shah J, Mukaetova-Ladinska EB, Hosseini AA. Memory impairment in Amyloidbeta-status Alzheimer's disease is associated with a reduction in CA1 and dentate gyrus volume: In vivo MRI at 7T. Neuroimage. 2024 Apr 15;292:120607. doi: 10.1016/j.neuroimage.2024.120607. Epub 2024 Apr 12. PMID 38614372